CLINICAL TRIAL: NCT04233125
Title: A Randomized Controlled Trial of Core Decompression With or Without Cement Packing for Osteonecrosis of the Femoral Head - Long Term Results
Brief Title: Core Decompression With or Without Cement Packing for ONFH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9604M11032
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Osteonecrosis
Keywords: Femoral Head; Hip; Core Decompression; Polymethlymethacrylate; Cement; Progression; Survival
MeSH Terms: conditions — Osteonecrosis; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Decompression (CD) Only (Active Comparator): Participants in this group receive standard care
  Interventions: Procedure: Core Decompression
- Added Polymethylmethacrylate (PMMA) (Experimental): Participants in this group receive standard care with an additional treatment
  Interventions: Procedure: Core Decompression; Procedure: PMMA augmentation

INTERVENTIONS:
Procedure: Core Decompression — Core Decompression
Procedure: PMMA augmentation — Polymethylmethacrylate (PMMA) augmentation
  Arms: Added Polymethylmethacrylate (PMMA)

SUMMARY:
Osteonecrosis of the femoral head (ONFH) is difficult to treat as collapse frequently occurs after core decompression (CD). This may be due to the failure to provide structural support during revascularization and healing. Reports of polymethylmethacrylate (PMMA) packing of the femoral head after CD for ONFH have noted favorable results. This study was undertaken to determine whether the addition of PMMA packing to CD provides any benefit to progression-free survival (PFS) and conversion to total hip arthroplasty-free survival (CFS). Secondary objectives were to assess for differences in functional outcomes and predictive factors for progression of the disease.

DETAILED DESCRIPTION:
A prospective randomized controlled trial comparing the results of CD vs. CD + PMMA packing in pre-collapse ONFH was set up.

Consecutive symptomatic patients aged >14 years with Association Research Circulation Osseous (ARCO) Stage I and II ONFH diagnosed using MRI and radiographic imaging were enrolled in this study.

Exclusion criteria were pre-existing collapse, sub-chondral fracture or degenerative changes of the hip.

After obtaining informed written consent, patients are asked to complete the Harris Hip Score (HHS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and a health status questionnaire Short Form-36 (SF-36).

The femoral heads enrolled into the study are randomized using a computer-generated card draw system to one of following: core decompression (CD) or core decompression with PMMA cement packing (CD + PMMA).

Allocation concealment was practiced with the use of opaque envelopes. Patients with bilateral involvement who had been randomized to one treatment modality for one femoral head were automatically selected to receive the other treatment modality for the contralateral femoral head.

Blinding of either surgeon or patient is impossible.

The patients were followed up after surgery every 3-4 months for the first 2 years after which the patients were seen annually. Completed questionnaires and radiographs were obtained at each visit.

Statistical Analysis The date of index procedure (CD or CD + PMMA) was used as start date for the purpose of statistical analysis. Progression Free Survival was defined as the time to radiographic progression and Conversion Free Survival (CFS) as the time to a THA. In case of patients who did not have radiographic progression, the date of their last follow up or death was used for the analysis. The SAS software will be used for all the analyses. The Log rank and Gerhan-Wilcoxon tests were used to compare Kaplan-Meier survival curves for the time from the date of the index procedure to radiographic progression (subchondral collapse) or conversion to THA for separate groupings based on age at index procedure (<40 , >40 yrs), smoking (Y/N), location (central, medial, lateral), percent involvement (<15% [mild], 15% to 30% [moderate], or >30% [severe]), index of necrotic extent (<40 or >40), and modified index of necrotic extent (<40 or >40). Whenever factors were found to affect the survival curves mainly in the initial year the Gerhan-Wilcoxon test was used as the test of significance. The Kaplan-Meier curves were also compared for the main cohorts of CD vs. CD + PMMA. Cox proportional hazards regression was used to compare factors (age, smoking, location, percent involvement, index of necrotic extent, and modified index of necrotic extent) with regards to their ability to predict the time to progression or revision to THA. Mixed multilevel regression modeling was used to test for group differences in the change in self-rated health survey scores over time from baseline over the post-operative period. The hierarchical linear modeling approach has a number of advantages over traditional repeated measures approaches for modeling change over time, including allowance for missing data and for varying measurement times across subjects. Separate models were generated for SF-36, Harris Hip Score and WOMAC scores over two-year and over 5-year post-operative time periods.

ELIGIBILITY:
Inclusion Criteria:

* Association Research Circulation Osseous (ARCO) Stage I and II ONFH diagnosed using MRI and radiographic imaging

Exclusion Criteria:

* pre-existing collapse, subchondral fracture or degenerative changes of the hip

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2005-01-01 (Actual); Study Completion 2008-01-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 5 years
  Progression Free Survival (PFS) is defined as the length of time (reported in months) following surgery that participants have no signs of radiographic progression of femoral head osteonecrosis. Radiographic progression is defined as any degree of flattening or loss of spherical contour of the femoral head as detected on the radiographs or MRI. Appearance of a subchondral fracture (crescent sign) on radiographs or MRI was also considered a sign of progression.

SECONDARY OUTCOMES:
Conversion Free Survival (CFS) | 5 years
  Conversion Free Survival (CFS) is defined as the length of time (reported in months) following surgery that participants are able to live without surgical conversion to total hip arthroplasty (THA).
Mean Harris Hip Score (HHS) | baseline, 2 years post surgery, 5 years post surgery
  The Harris Hip Score (HHS) is a clinician-based instrument with 4 sub-scales measuring pain severity (44 points), function (47 points), absence of deformity (4 points), and range of motion (5 points). Total score is calculated as a sum of 4 sub-scale scores and ranges from 0-100 with higher scores representing less dysfunction. Three time points will be reported.
Change in Harris Hip Score (HHS) | baseline, 2 years post surgery
  The Harris Hip Score (HHS) is a clinician-based instrument with 4 sub-scales measuring pain severity (44 points), function (47 points), absence of deformity (4 points), and range of motion (5 points). Total score is calculated as a sum of 4 sub-scale scores and ranges from 0-100 with higher scores representing less dysfunction.
Mean Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline, 2 years post surgery, 5 years post surgery
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items), stiffness (2 items), and physical function (17 items). Items are rated on a Likert scale of 0 (extreme) to 4 (none). Raw sub-scale scores are normalized by multiplying each score by 100/96. Total scores are a sum of the normalized sub-scales scores and range 0-100, with higher scores indicating better functioning. Three time points will be reported.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline, 2 years post surgery
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items), stiffness (2 items), and physical function (17 items). Items are rated on a Likert scale of 0 (extreme) to 4 (none). Raw sub-scale scores are normalized by multiplying each score by 100/96. Total scores are a sum of the normalized sub-scales scores and range 0-100, with higher scores indicating better functioning.
Mean Short Form-36 (SF-36) | baseline, 2 years post surgery, 5 years post surgery
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health, containing 8 scaled sub-scores: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each sub-scale score is calculated as the weighted sum of the questions in that section, then directly transformed into a 0-100 score using a scoring algorithm. The SF-36 also produces two summary scores, physical component summary and the mental component summary. Lower scores indicated greater disability. Three time points will be reported.
Change in Short Form-36 (SF-36) | baseline, 2 years post surgery
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health, containing 8 scaled sub-scores: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each sub-scale score is calculated as the weighted sum of the questions in that section, then directly transformed into a 0-100 score using a scoring algorithm. The SF-36 also produces two summary scores, physical component summary and the mental component summary. Lower scores indicated greater disability.

IPD SHARING:
Plan to Share IPD: No